CLINICAL TRIAL: NCT05553301
Title: Safety and Immunogenicity of Quadrivalent Influenza mRNA Vaccine MRT5407 in Adults Aged 18 Years and Older
Brief Title: Safety and Immunogenicity of Quadrivalent Influenza mRNA Vaccine MRT5407 in Adult Participants18 Years of Age and Older
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAV00002; U1111-1271-1302 (Registry Identifier: ICTRP)
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Influenza Immunization
MeSH Terms: conditions — Influenza, Human | interventions — Vaccines; Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Sentinel Cohort: Open label
  Main Cohort:
  * Open label (Sponsor, except laboratory testing personnel)
  * Blinded (Sites, except for those preparing/administering study intervention)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a parallel-group prevention study with up to 5 arms that will be blinded to participants, investigators / sub-investigators, outcomes assessors, and laboratory personnel (with the exception of the sentinel safety portion of the study, which will be open-label). The Sponsor study staff will be unblinded (except laboratory testing personnel).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Group 1: Quadrivalent Influenza mRNA Vaccine MRT5407 dose level 1 (Experimental): participants will receive a single dose of QIV mRNA vaccine (dose level 1)
  Interventions: Biological: Quadrivalent Influenza mRNA Vaccine MRT5407
- Group 2: Quadrivalent Influenza mRNA Vaccine MRT5407 dose level 2 (Experimental): participants will receive a single dose of QIV mRNA vaccine (dose level 2)
  Interventions: Biological: Quadrivalent Influenza mRNA Vaccine MRT5407
- Group 3: RIV4 (Active Comparator): participants will receive a single dose of RIV4 vaccine
  Interventions: Biological: Quadrivalent Recombinant Influenza Vaccine
- Group 4: QIV-SD (Active Comparator): participants will receive a single dose of QIV-SD vaccine
  Interventions: Biological: Quadrivalent Influenza Standard Dose Vaccine
- Group 5: QIV-HD (Active Comparator): participants will receive a single dose of QIV -HD vaccine (for elderly only)
  Interventions: Biological: Quadrivalent Influenza High-Dose Vaccine

INTERVENTIONS:
Biological: Quadrivalent Influenza mRNA Vaccine MRT5407 — Pharmaceutical Form: Liquid frozen solution in a vial
  Route of Administration: Intramuscular Injection
  Arms: Group 1: Quadrivalent Influenza mRNA Vaccine MRT5407 dose level 1; Group 2: Quadrivalent Influenza mRNA Vaccine MRT5407 dose level 2
Biological: Quadrivalent Recombinant Influenza Vaccine — Pharmaceutical Form: Liquid frozen solution in a vial
  Route of Administration: Intramuscular Injection
  Other Names: Flublok Quadrivalent®
  Arms: Group 3: RIV4
Biological: Quadrivalent Influenza Standard Dose Vaccine — Pharmaceutical Form: Liquid suspension for injection in pre-filled syringe
  Route of Administration: Intramuscular Injection
  Other Names: Fluzone Qudrivalent®
  Arms: Group 4: QIV-SD
Biological: Quadrivalent Influenza High-Dose Vaccine — Pharmaceutical Form: Liquid suspension for injection in pre-filled syringe
  Route of Administration: Intramuscular Injection
  Other Names: Fluzone High-Dose Quadrivalent®
  Arms: Group 5: QIV-HD

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of a single intramuscular (IM) injection of up to 2 dose levels of Quadrivalent Influenza messenger ribonucleic acid (mRNA) Vaccine MRT5407 compared to an active control (QIV standard-dose (SD), QIV high-dose (HD) [adults ≥ 65 years of age only], or quadrivalent recombinant influenza vaccine (RIV4)) in adults 18 years of age and older.

DETAILED DESCRIPTION:
Study duration is approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years on the day of inclusion
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year, or surgically sterile OR
  * Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 12 weeks after study intervention administration.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Previous history of myocarditis, pericarditis, and / or myopericarditis
* Self-reported thrombocytopenia, contraindicating Intramuscular vaccination based on Investigator's judgment
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating Intramuscular vaccination based on Investigator's judgment
* Moderate or severe acute illness / infection (according to Investigator's judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of vaccination. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Self-reported or documented seropositivity for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus
* Receipt of any mRNA vaccine/product in the 2 months preceding study intervention administration

NOTE: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with immediate adverse events (AEs) | Within 30 minutes after injection
  Unsolicited systemic AEs that occur within 30 minutes after vaccination
Number of participants with solicited injection site and systemic reactions | Up to 7 days after injection
  Adverse reactions pre-listed in the protocol and case report form (CRF) Injection site reactions: pain, redness, swelling, hardening, bruising Systemic reactions: fever, headache, malaise, myalgia, arthralgia, chills
Number of participants with unsolicited AEs | Up to 28 days after injection
  AEs that do not fulfill the conditions of solicited reactions
Number of participants with medically attended adverse events (MAAE)s | Up to 28 days after injection
  AEs with a new onset or a worsening of a condition that prompts the participant or participant to seek unplanned medical advice at a physician's office or Emergency Department
Number of participants with serious adverse events (SAEs) | From Day one to Day 366
  SAEs reported throughout the study
Number of participants with out-of-range biological test results | Up to 8 days after injection
  Out-of-range biological test results (including shift from baseline values)
Individual Hemagglutination inhibition (HAI) titer | At Day 1 and Day 29
  Antibody titers are expressed as GMTs at baseline and post-baseline
Percentage of participants with detectable antibody HAI titers greater than or equal to (≥) 10 [1/dil] | At Day 1 and Day 29
Individual HAI titer ratio | At Day 1 and Day 29
  Ratios of antibody titers measured by HAI in each group before and after vaccination
Number of participants archiving HAI seroconversion against Antigens | At Day 1 and Day 29
  Number of participants with titer < 10 [1/dil] at Day 1 and post-vaccination titer ≥ 40 [1/dil] at Day 29, or titer ≥ 10 [1/dil] at Day 1 and a ≥ 4-fold-rise in titer [1/dil] at Day 29
Percentage of participants with antibody HAI titers greater than or equal to (≥) 40 [1/dil] | At Day 29
Percentage of participants with 2-fold and 4-fold rise in HAI titers | At Day 1 and Day 29

SECONDARY OUTCOMES:
Neutralizing Ab titers | At Day 1 and Day 29
  Neutralizing Ab titers expressed as GMTs
Individual neutralizing antibodies titer ratio | At Day 1 and Day 29
Percentage of participants with 2-fold and 4-fold increase in neutralizing titers | At Day 1 and Day 29
Individual HAI Ab titer ratio | Day 1, Day 91, Day 181 and Day 366
Percentage of participants with antibody HAI titers greater than or equal to (≥) 40 [1/dil] | At Day 91, Day 181 and Day 366
Individual neutralizing Ab titer ratio | Day 1, Day 91, Day 181 and Day 366

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (25):
- United States (23):
  - Peninsula Research Associates Site Number : 8400025, Rolling Hills Estates, California
  - Optimal Research Site Number : 8400059, San Diego, California
  - California Research Foundation Site Number : 8400008, San Diego, California
  - Accel Clinical Research-Deland Clinical Research Unit Site Number : 8400052, DeLand, Florida
  - SIMEDHealth, LLC Site Number : 8400024, Gainesville, Florida
  - Indago Research and Health Center Site Number : 8400014, Hialeah, Florida
  - Cenexel Research Centers of America Site Number : 8400048, Hollywood, Florida
  - Dade Research Center Site Number : 8400011, Miami, Florida
  - Suncoast Research Group, LLC Site Number : 8400038, Miami, Florida
  - Florida International Research Center Site Number : 8400051, Miami, Florida
  - Palm Beach Research Center Site Number : 8400020, West Palm Beach, Florida
  - DM Clinical Research Site Number : 8400032, Melrose Park, Illinois
  - DM Clinical Research - Chicago Site Number : 8400028, River Forest, Illinois
  - Brengle Family Medicine Site Number : 8400005, Indianapolis, Indiana
  - AMR Lexington Site Number : 8400054, Lexington, Kentucky
  - AMR Kansas City Site Number : 8400006, Kansas City, Missouri
  - Velocity Clinical Research Site Number : 8400003, Omaha, Nebraska
  - Coastal Carolina Research Center - N Charleston Site Number : 8400010, North Charleston, South Carolina
  - AMR Knoxville Site Number : 8400046, Knoxville, Tennessee
  - Elligo Health Research Site Number : 8400056, Austin, Texas
  - Sun Research Institute Site Number : 8400030, San Antonio, Texas
  - Clinical Trials of Texas, Inc. Site Number : 8400026, San Antonio, Texas
  - DM Clinical Research - Sugar Land Site Number : 8400031, Sugar Land, Texas
- Puerto Rico (2):
  - Investigational Site Number : 6300003, Barrio Sabana
  - Investigational Site Number : 6300002, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org